CLINICAL TRIAL: NCT03202667
Title: Effects of the SGLT2-inhibitor Empagliflozin on Patients With Chronic SIADH - the SANDx Study
Acronym: SANDx
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-00701
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: SIAD - Syndrome of Inappropriate Antidiuresis; Hyponatremia
Keywords: SGLT2-inhibitor; Treatment
MeSH Terms: conditions — Inappropriate ADH Syndrome; Hyponatremia | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin (Active Comparator): Treatment with empagliflozin 25mg tablets once daily for 28 days
  Interventions: Drug: Empagliflozin 25mg
- Placebo (Placebo Comparator): Treatment with Placebo tablets once daily for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 25mg — Treatment with empagliflozin 25mg once daily for 28 days
  Arms: Empagliflozin
Drug: Placebo — Treatment with Placebo oral tablet once daily for 28 days
  Arms: Placebo

SUMMARY:
Syndrome of inappropriate antidiuresis (SIADH) is characterized by an imbalance of antidiuretic vasopressin (AVP) secretion. The impaired AVP regulation leads to water retention and secondary natriuresis and is a common cause for hyponatremia.

Especially chronic (>72h) SIADH is difficult to treat as standard therapeutic options (water restriction, urea, salt tablets) often do not succeed in correction of hyponatremia, making additional therapy necessary.

Empagliflozin is a sodium glucose co-transporter 2 (SGLT2)-inhibitor, which is a well-tolerated treatment option for type 2 diabetes mellitus. The inhibition of SGLT2 in the proximal tubule leads to renal excretion of glucose with subsequent osmotic diuresis. This mechanism could result in a therapeutic effect in patients with chronic SIADH, as it resembles the aquaretic effect of urea.

The aim of this study is to evaluate whether empagliflozin has an effect on the serum sodium levels of patients with chronic SIADH.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (age ≥ 18 years) with hyponatremia (<133mmol/l) due to chronic (>72h) SIADH defined as

* serum osmolality <275mosm/kg
* urine osmolality >100mosm/kg
* urine sodium >30mmol/l

Exclusion Criteria:

* acute (<72h) or transient hyponatremia
* severe symptomatic hyponatremia in need of hospital treatment
* diabetes mellitus type 1
* uncontrolled hypothyroidism
* uncontrolled adrenal insufficiency
* renal impairment (GFR <45ml/min)
* cardiac failure
* symptomatic liver disease / severe hepatic impairment (ALAT / aspartate transaminase (ASAT) > 3x upper limit)
* treatment with SGLT 2 inhibitors, lithium chloride, urea or glitazone
* severe immunosuppression
* pregnancy or breastfeeding
* palliative situation (end of life care)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Change in Serum Sodium concentration | 28 days
  Difference in serum sodium concentration in mmol/l after 28 days of treatment

SECONDARY OUTCOMES:
Change in Serum sodium concentration | 21 days
  Serum sodium concentration 1, 2 and 3 weeks of treatment
Change in Serum electrolytes | 28 days
  Serum electrolytes after 1, 2, 3 and 4 weeks of treatment
Urinary electrolytes | 7 days
  Urinary electrolytes after 1 week of treatment
Urinary electrolytes | 14 days
  Urinary electrolytes after 2 weeks of treatment
Urinary electrolytes | 21 days
  Urinary electrolytes after 3 weeks of treatment
Urinary electrolytes | 28 days
  Urinary electrolytes after 4 weeks of treatment
Serum osmolality | 7 days
  Serum osmolality after 1 week of treatment
Serum osmolality | 14 days
  Serum osmolality after 2 weeks of treatment
Serum osmolality | 21 days
  Serum osmolality after 3 weeks of treatment
Serum osmolality | 28 days
  Serum osmolality after 4 weeks of treatment
Urinary osmolality | 7 days
  Urinary osmolality after 1 week of treatment
Urinary osmolality | 14 days
  Urinary osmolality after 2 weeks of treatment
Urinary osmolality | 21 days
  Urinary osmolality after3 weeks of treatment
Urinary osmolality | 28 days
  Urinary osmolality after 4 weeks of treatment
Serum glucose | 7 days
  Serum glucose after 1 week of treatment
Serum glucose | 14 days
  Serum glucose after 2 weeks of treatment
Serum glucose | 21 days
  Serum glucose after 3 weeks of treatment
Serum glucose | 28 days
  Serum glucose after 4 weeks of treatment
Urinary glucose | 7 days
  Urinary glucose after 1 week of treatment
Urinary glucose | 14 days
  Urinary glucose after 2 weeks of treatment
Urinary glucose | 21 days
  Urinary glucose after 3 weeks of treatment
Urinary glucose | 28 days
  Urinary glucose after 4 weeks of treatment
Copeptin | 7 days
  Plasma copeptin after 1 week of treatment
Copeptin | 14 days
  Plasma copeptin after 2 weeks of treatment
Copeptin | 21 days
  Plasma copeptin after3 weeks of treatment
Copeptin | 28 days
  Plasma copeptin after 4 weeks of treatment
Aldosterone | 7 days
  Plasma aldosterone after 1 week of treatment
Aldosterone | 14 days
  Plasma aldosterone after 2 weeks of treatment
Aldosterone | 21 days
  Plasma aldosterone after 3 weeks of treatment
Aldosterone | 28 days
  Plasma aldosterone after 4 weeks of treatment
Renin | 7 days
  Plasma renin after 1 week of treatment
Renin | 14 days
  Plasma renin after 2 weeks of treatment
Renin | 21 days
  Plasma renin after 3 weeks of treatment
Renin | 28 days
  Plasma renin after 4 weeks of treatment
MR-proANP | 7 days
  Plasma MR-proANP after 1 week of treatment
MR-proANP | 14 days
  Plasma MR-proANP after 2 weeks of treatment
MR-proANP | 21 days
  Plasma MR-proANP after 3 weeks of treatment
MR-proANP | 28 days
  Plasma MR-proANP after 4 weeks of treatment
N terminal (NT)-proBNP | 7 days
  Plasma NT-proBNP after 1 week of treatment
NT-proBNP | 14 days
  Plasma NT-proBNP after 2 weeks of treatment
NT-proBNP | 21 days
  Plasma NT-proBNP after 3 weeks of treatment
NT-proBNP | 28 days
  Plasma NT-proBNP after 4 weeks of treatment
P1NP | 7 days
  Plasma P1NP after 1 week of treatment
P1NP | 14 days
  Plasma P1NP after 2 weeks of treatment
P1NP | 21 days
  Plasma P1NP after 3 weeks of treatment
P1NP | 28 days
  Plasma P1NP after 4 weeks of treatment
CTx | 7 days
  Plasma CTx after 1 week of treatment
CTx | 14 days
  Plasma CTx after 2 weeks of treatment
CTx | 21 days
  Plasma CTx after 3 weeks of treatment
CTx | 28 days
  Plasma CTx after 4 weeks of treatment
Osteocalcin | 7 days
  Plasma Osteocalcin after 1 week of treatment
Osteocalcin | 14 days
  Plasma Osteocalcin after 2 weeks of treatment
Osteocalcin | 21 days
  Plasma Osteocalcin after 3 weeks of treatment
Osteocalcin | 28 days
  Plasma Osteocalcin after 4 weeks of treatment
General well being (assessed by VAS) | 28 days
  General well being after 1, 2, 3 and 4 weeks of treatment
Headache (assessed by VAS) | 28 days
  Headache after 1, 2, 3 and 4 weeks of treatment
Vertigo (assessed by VAS) | 28 days
  vertigo after 1, 2, 3 and 4 weeks of treatment
Nausea (assessed by VAS) | 28 days
  Nausea after 1, 2, 3 and 4 weeks of treatment
Malaise (assessed by VAS) | 28 days
  Malaise after 1, 2, 3 and 4 weeks of treatment
Body weight (kg) | 28 days
  Body weight after 1, 2, 3 and 4 weeks of treatment
Blood pressure (mmHg) | 28 days
  Blood pressure after 1, 2, 3 and 4 weeks of treatment
Heart rate (bpm) | 28 days
  Heart rate after 1, 2, 3 and 4 weeks of treatment
Neurocognitive function (assessed by MOCA) | 28 days
  change in Neurocognitive function (baseline versus after 4 weeks of Treatment)
Muscle strength (measured by grip strength test) | 28 days
  Change in Muscle strength (baseline vs after 4 weeks of Treatment)
Gait Dynamics (measured by gait Analysis) | 28 days
  Gait dynamics baseline vs after 4 weeks of treatment
Hemodynamic Parameters (measured by thoracic electrical bioimpedance) | 28 days
  Hemodynamic parameters baseline vs after 4 weeks of treatment
Body fluid volume (measured by bioimpedance spectroscopy) | 28 days
  Body fluid volume baseline vs after 4 weeks of treatment
Amount of Fluid intake in ml | 28 days
  Fluid intake after 1, 2, 3 and 4 weeks of treatment
Number of Falls | 30 days
  Rate of falls during observation phase
number of Fractures | 30 days
  Rate of fractures during observation phase
number of Hospital admissions | 30 days
  Rate of Hospital admissions during observation phase
Hyponatremia recurrence | 30 days
  Rate of hyponatremia recurrence during 30day follow up

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. Dr. MD, Study Director — University Hopsital Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Monnerat S, Refardt J, Potasso L, Meier C, Christ-Crain M. An Increase in Plasma Sodium Levels Is Associated With an Increase in Osteoblast Function in Chronic SIAD. J Clin Endocrinol Metab. 2023 Sep 18;108(10):e1027-e1033. doi: 10.1210/clinem/dgad238. PMID 37098131
- [Derived] Refardt J, Imber C, Nobbenhuis R, Sailer CO, Haslbauer A, Monnerat S, Bathelt C, Vogt DR, Berres M, Winzeler B, Bridenbaugh SA, Christ-Crain M. Treatment Effect of the SGLT2 Inhibitor Empagliflozin on Chronic Syndrome of Inappropriate Antidiuresis: Results of a Randomized, Double-Blind, Placebo-Controlled, Crossover Trial. J Am Soc Nephrol. 2023 Feb 1;34(2):322-332. doi: 10.1681/ASN.2022050623. Epub 2022 Nov 17. PMID 36396331